CLINICAL TRIAL: NCT03563131
Title: Tibial and Femoral Components Migration and Adaptive Bone Remodeling After Insertion of Persona® Total Knee Arthroplasty. A RCT Using RSA and DEXA Analysis for Evaluation of Uncemented With Trabecular Metal Surface vs. Cemented Fixation
Brief Title: Tibial and Femoral Components Migration and Adaptive Bone Remodeling After Insertion of Persona® TKA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Gentofte Hospital, Denmark (Unknown)
Responsible Party: Principal Investigator, Müjgan Yilmaz, Medical Doctor,Research Fellow, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PERSONA-RH-18
Record Dates: First submitted 2018-06-08; First posted 2018-06-20 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Osteo Arthritis Knee
Keywords: Osteoarthritis; Knee; Arthroplasties
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uncemented Persona® total knee arthroplasty (Active Comparator): Uncemented TM Zimmer Persona® TKA. It is a relatively new implant that is now in routine clinical use. Implants are approved by FDA and CE marked. Patella will be resurfaced with the cemented Zimmer 3-Peg All Polyethylene Patella.
  Interventions: Device: Persona® total knee arthroplasty
- Cemented Persona® total knee arthroplasty (Active Comparator): Cemented Zimmer Persona® TKA. It is a relatively new implant that is now in routine clinical use. Implants are approved by FDA and CE marked. Patella will be resurfaced with the cemented Zimmer 3-Peg All Polyethylene Patella.
  Interventions: Device: Persona® total knee arthroplasty

INTERVENTIONS:
Device: Persona® total knee arthroplasty — Insertion of the cemented or uncemented Persona® total knee arthroplasty

SUMMARY:
The purpose of this study:

In a prospective randomized study with 2 years of follow-up we want to compare the migration of the uncemented trabecular metal (TM) versus the cemented tibial and femoral components of the new Persona® total knee arthroplasty (TKA) assessed by model based radiostereometric analysis (MB-RSA). Also, we want to compare the adaptive bone remodeling induced by the uncemented TM versus the cemented tibial and femoral components of the new Persona® TKA assessed by dual energy-X-ray (DEXA). Data generated for both above mentioned, will be also compared with historical RSA and DEXA data for the NexGen TKA using TM tibia modular and monoblock.

DETAILED DESCRIPTION:
Detailed Description: Main Hypothesis:

1. The uncemented TM Zimmer Persona® TKA will have migration on the same level as the cemented Zimmer Persona® TKA.
2. The uncemented TM Zimmer Persona® TKA will have less loss of BMD compared to the cemented version of the implant.

Material and Methods:

A prospective randomized study where the patients scheduled for TKA are randomized to receive tibial and femoral components with two different fixation modes:

Group A: an uncemented TM Zimmer Persona® TKA (uncemented tibia and femur components).

Group B: a cemented Zimmer Persona® TKA (cemented tibia and femur components). Operation: Operation Planning of the operations are performed based upon standing knee X-rays (not involving the ankle and hip joint) and no preoperative templating is performed. The operations are performed at the Department of Orthopedic Surgery, Gentofte Hospital by three experienced TKA surgeons that will be included in the research group. All patellas will be resurfaced with a cemented all polyethylene patella component. During surgery the patients participating in the study will be prepared for MB-RSA by insertion of a minimum of 6 Tantalum markers (0.8 mm) in the bone of the proximal tibia and 6 markers in the distal femur.

Intravenous antibiotics (1.5g Cefuroxim) are administered three times during the first day and night of surgery and low molecular weight heparin is administered for prevention of deep venous thrombosis and pulmonary embolism. Local analgesics (Naropin ®, Toradol ®) are injected in the knee joint and in the soft tissue around the knee during surgery. Physiotherapy begins on the day of surgery and the patients will be mobilized with full weight-bearing using crutches.

Research plan

1. Clinical examination (n=60): preoperatively and with follow-up after 1 and 2 years with evaluation of the knee function using the Knee Society's Knee Scoring System.
2. Patient-reported outcome measurements (n=60). Obtained preoperatively and after 1 and 2 years using the Oxford knee score.
3. Conventional X-rays (n=60) are obtained preoperatively (standing knee X-rays (not involving the ankle and hip joint)), with classification of the degree of arthrosis estimating the Ahlbäck score. X-rays are also obtained postoperatively before the patients are discharged and after 1 year and 2 years with the aim of evaluating knee alignment, and development of osteolytic lesions.
4. CT-scans (n=60) 3 months postoperatively for measurements of hip-knee-ankle (HKA) angle, and component slope, rotation, and size matching.
5. Special X-rays suitable for MB-RSA measurements (n=60) of migration of the tibial and femoral components is performed within the first week after the operation and after 3, 6, 12, and 24 months. The precision of the RSA measurements is estimated from double examinations in 12 patients of the study. RSA X-rays will be performed using a biplane RSA arrangement with a 90° angle between the two X-ray tubes (Calibration cage 21; Tilly Medical Products AB, Lund, Sweden) and analysis of X-rays will be performed by the MB-RSA commercial software (RSAcore, Department of Orthopedics, Leiden University Medical Center, Leiden, The Netherlands), available at the Skaane University Hospital, Lund, Sweden. The manufacturer (Zimmer Biomet) will provide the CAD models.
6. DEXA analysis of the adaptive changes in BMD of the periprosthetic bone of the distal femur and proximal tibia. DEXA analysis will be performed preoperatively of the distal femur (lateral projection) and proximal tibia (coronal projection) as baseline, then again within the first postoperative week and subsequently at 3 months, 6 months, 1 year, and 2 years. The precision of the BMD measurements of the proximal tibia and distal femur will be estimated from double measurements of patients (n=12) included in the study.

Calculation of sample size MB-RSA There exist only three previously published studies measuring femoral component migration. In all studies the marker-based RSA technique was used, and none of them presented results with mean and standard deviation (SD). However, one study gave the results as mean MTPM, and we chose the mean MTPM after 2 years of follow-up (0.88 mm for cemented components) as our primary effect parameter, used in the sample size calculation. The rationale for using MTPM two years postoperatively, is because it has been shown to be the best predictor for later aseptic loosening of the tibial component after primary TKA. SD was estimated from the most recently published study using MB-RSA for evaluation of cemented tibial component migration. In that study, the mean (+/- SD) MTPM after 2 years of follow-up was 0.47 (+/- 0.16) and 0.45 (+/-0.21) in the two study groups. Since the level of MTPM of the tibial components was substantially lower than seen for the above mentioned femoral components. We adjusted the SD in the sample size calculation to constitute the same percentages of the mean values as in the tibial component MB-RSA study by Ejaz et al. (2015). Since the previously published studies measuring femoral component migration did not find any statistically significant difference between cemented and uncemneted fixation we selected a relatively low minimum relevant difference (MIREDIF).

Using:

Type I error = 5% Statistical power = 85 % MIREDIF 0.3 mm SD = 0.35 mm Sample size calculation resulted in a sample size of n = 24 in each group. In the study we have planned to include and randomize (block-randomization with 10 in each block) a total of 60 patients. This will secure a high statistical power even if some of the participants should drop out during the study.

DEXA

The data for the sample size calculations were obtained from new DEXA data for our own research group: data from a study evaluating the adaptive bone remodeling around the Vanguard® uncemented porous-coated femoral component with one year of follow-up. Using one-year follow-up data could be justified because the decrease in BMD seen beyond the first postoperative year is very limited in most studies. We considered a difference of 8% between groups to be a clinically relevant difference that we wanted to be able to detect with a high statistical power:

Using:

Type I error = 5% Statistical power = 90 % MIREDIF 8% SD = 8.4% Sample size calculation resulted in a sample size of n = 25 in each group.

In the study we have planned to include and randomize (block-randomization with 10 in each block) a total of 60 patients. This will secure a high statistical power even if some of the participants should drop out during the study.

Ethical considerations We do not expect that the patients participating in the study will experience any special side effects or complications related to the use of the two TKAs.

There has not been performed any fundamental changes in implant design compared to other types of standard TKAs and the implant fixation modes (cemented or uncemented with a TM ingrowth surface) are well known and in wide spread use.

Radiation dose to the patients from MB-RSA X-rays and DEXA is relatively low compared with many conventional X-ray examinations.The total accumulated radiation dose to a patient participating in all examinations during the study is estimated to be approximately 2 mSv.

Tantalum has been used for more than 50 years and is a very biocompatible material without any tendency to corrosion.Tantalum beads for RSA have been used in several clinical studies for more than 20 years. More than 20.000 beads have been implanted in more than 2.000 patients and no side effects from Tantalum beads have been observed.

This investigation will be performed in accordance with the principles of the Helsinki Declaration, and all patients will receive both oral and written information before informed consent to participate is obtained. At any time being the patient will be able to cancel participation (also without any explanation) in this investigation. The patient will receive the best possible treatment in any circumstances. The study will not be started until approval from the Scientific Ethical Committee of the Capital Region of Denmark and the Danish Data Protection Agency has been obtained, and it will be registered at clinicaltrials.gov.

Risks and inconveniences:This investigation will not add to the general risks of getting TKA. Patients participating must accept some inconvenience in terms of additional examinations and hence transportation to and from the hospitals.

Adverse events: All adverse events will be recorded in the CRF and will include details concerning the nature, onset, duration, severity, relationship to the device and relationship to the operative procedure and outcome. The affected patient(s) will be questioned about any adverse event(s) at each subsequent follow-up visit.

Patients experiencing adverse events will be relevantly monitored by clinical assessment and lab examinations decided by the treating physician. All adverse events will be monitored until recovery or stabilization.

Information and consent Patients who are planned to receive a TKA (and fits within the inclusion and exclusion criteria of the study) at Gentofte Hospital will be informed about the trial in the preoperative interview. In addition to the oral information provided, the patients will be given written information. This conversation will take place in an enclosed space without distractions or interruptions. The patient will receive adequate verbal and written information about the purposes, processes, potential benefits and risks including possible side effects. Investigator will ensure all patients have read and understood the information and consent form. Patients will be informed that they are entitled to consideration before consent is given. The subjects will also be informed that it is voluntary and that they at any time may withdraw from the trial. It is the investigator's responsibility to ensure the above.

There will be obtained written informed consent from all subjects before enrollment, and a copy of the information and consent form will be given to the subjects.Existing legislations made by the Scientific Ethical Committee regarding informed consent will be followed.

Data protection All information will be kept confidential, and all data handled according the guidelines of the Danish Data Protection agency. The persons involved in this trial are obliged to professional secrecy. The investigator will maintain a list of identification of all enrolled patients. This list will contain the patients' full names and dates of birth (including social security numbers (CPR-numbers)).

Collected data will be recorded in a case report form (CRF). CRFs and the medical records will be made available to third parties according to Danish law. Patients will be informed in writing that the results will be stored and analyzed in a computer which preserve patients' anonymity and that the local laws regarding personal data will be complied.

Patients will also receive written information concerning the possibility of audit from the public authorities, and patients will be informed that the GCP unit of Copenhagen University Hospital likewise is granted access.

Investigator ensures that the project will follow the rules of Good Clinical Practice

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthrosis of the knee with indication for a TKA.
* Age between 40 and 70 years.

Exclusion Criteria:

* If a standard cruciate retaining implants cannot be used due to e.g. severe malalignment/deformity or instability.
* Diseases affecting the bone metabolism (severe osteoporosis, Pagets disease, hyperparathyreoidism etc.).
* Patients estimated not to be able to understand the "Information to patients" papers or do not want to participate in the study.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Migration | 2 years
  The differences between the cemented and uncemented implants are evaluated by measurements of migration of the stem assesed by Radiosteriometric analysis (RSA), measuring the migration by the MB-RSA Commercial software.

SECONDARY OUTCOMES:
Adaptive bone remodelling | 2 years
  The difference of the cemented and uncemented implants are evaluated by measurements of the adaptive bone remodeling of the periprostetic area assesed by dual energy X-ray absorptiometry (DXA), that measures body mass density (BMD)

OTHER OUTCOMES:
Knee function assessed with Knee Society Score | 2 years
  Knee function postoperatively assessed by the Knee Society's Knee Scoring System (an objective scoring system to rate the knee and patient's functional abilities such as walking and stair climbing. Max score: 100; Min score: below 60 )
Knee function assessed with Oxford Knee Score | 2 years
  Oxford Knee Score (a Patient Reported Outcome questionnaire developed to assess the patient's perspective of outcome following Total Knee Arthroplasty. Max score: 48; Min score 0)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Petersen, Professor, Study Director — Rigshospitalet, Denmark
Locations (1):
- Gentofte Hospital, Hellerup, Denmark